CLINICAL TRIAL: NCT04147871
Title: A Multicentre, Randomized, Controlled Versus Placebo, Double-blinded, 4 Parallel Arms, Dose-ranging Main Study, to Evaluate the Efficacy, Safety and Tolerability and Acceptability of Repeated Doses of ADV7103, After 7 Days of Treatment, in Patients With Cystinuria, and an Efficacy and Safety Exploratory Study in the Youngest Children.
Brief Title: Study Evaluating Patients With Cystinuria and Efficacy and Safety Exploratory Study in the Youngest Children
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unspecified business decision/strategic reason
Sponsor: Advicenne Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B12CS-B13CS
Record Dates: First submitted 2019-10-23; First posted 2019-11-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2023-05

CONDITIONS: Cystinuria
MeSH Terms: conditions — Cystinuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ADV7103 1.5 mEq/Kg/day (Active Comparator): Patients receive ADV7103 twice a day.
  Interventions: Drug: ADV7103
- ADV7103 3.0 mEq/Kg/day (Active Comparator): Patients receive ADV7103 twice a day.
  Interventions: Drug: ADV7103
- ADV7103 4.5 mEq/Kg/day (Active Comparator): Patients receive ADV7103 twice a day.
  Interventions: Drug: ADV7103
- Placebo (Placebo Comparator): Patients receive placebo twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADV7103 — Each dose of ADV7103 contains a fixed ratio of 1/3 of ADV7103-CK (potassium citrate) and 2/3 of ADV7103-BK (potassium bicarbonate) based on the mass of active substances.
  Arms: ADV7103 1.5 mEq/Kg/day; ADV7103 3.0 mEq/Kg/day; ADV7103 4.5 mEq/Kg/day
Drug: Placebo — Placebo is a combination of 2 mm green coated lactose granules and 2 mm white coated lactose granules.
  Each dose of placebo contains a fixed ratio of 1/3 of green granules and 2/3 of white granules.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, controlled versus placebo, double-blinded, 4 parallel arms, dose-ranging main study, to evaluate the efficacy, safety and tolerability, and acceptability of repeated doses of ADV7103, after 7 days of treatment, in patients with cystinuria, and an efficacy and safety exploratory study in the youngest children.

DETAILED DESCRIPTION:
The study will target enrolling at least 15 subjects in each of the following age groups: 6 months - 5 years (B13CS part only); 6-11 years; 12-17 years and adults>18. Subjects will be in the study for up to 7 weeks.

After screening and enrollment (up to 35 days), Eligible patients will be treated will alkalinizing treatment (SoC) at the well-adapted dose and regimen for 7 days. An in-patient visit is planned at the end of this period. The baseline evaluations, including urine pH and specific gravity, will be done during this inpatient visit, from Day -1 t0 to t24h. After this visit, patients are randomized in a balanced manner (1:1:1:1) to one of the 4 possible treatment arms, ADV7103 at a low dose, medium dose or high dose, or ADV7103 placebo. For patients in B13CS part, a period of titration is planned before the 7 days of treatment with ADV7103. No use of placebo in B13CS.

Controls of urine pH will be done at the patient's home with a pocket glass electrode pH-meter on fresh urines, at least twice a day: before the administration of ADV7103, in the morning at t0 and in the evening at t12h (12hrs after last ADV7103 intake and before the next dose).

Subjects will have the opportunity to subsequently enter a long-term, open-label extension.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient who has a diagnosis of cystinuria based on medical diagnosis (at least one previous orcurrent episode of calculus of cystine, and/or one previous or current episode of cystine crystalluria) or on genetic diagnosis (only for patients enrolled in B13CS study).

  2. Patient treated with an alkalising treatment at a well-adapted dose (defined as a daily dose deemed by the investigator aiming to maintain overtime urinary pH value ≥ 7.0 and/or compatible with an acceptable safety profile and/or patient's constraints or compliance).

  3. Patient who, when treated with a second line therapy (chelator agent), presents a disease status enabling interruption of the chelator agent during the course of the B12CS-B13CS research.

  4. Patient male or female, including child aged between 6 months and 17 years old and adult aged ≥ 18 years old up to 70 years old.

  5. For female patient of childbearing potential (defined by CTFG as fertile, following menarche until becoming post-menopausal unless permanently sterile*) a highly effective birth control method should be used until the end of study plus 36 hours after the last dose of IMP.

  6. Patient and/or parents or legal representative(s) who is(are) willing and able to participate in the study, to understand and to comply with study procedures for the entire length of the study.

  7. Patient or parents or legal representative(s) who has/have provided a signed written informed consent.

  8. Patient of ≤17 years of age for whom the assent has been collected or has been tried to be collected.

  9. Patient who is affiliated to a social health insurance system and/or in compliance with the recommendations of the national law in force relating to biomedical research.

Exclusion Criteria:

* 1. Patient treated with the second line therapy and who cannot stop cystine chelating agents (sulfhydryl compounds) during the B12CS-B13CS study.

  2. Patient who presents kalaemia > 5.0 mmol/L. 3. Patient who presents a moderate or severe renal impairment (estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2 according to Schwartz formula for the children and both MDRDs and CKD-EPI for adults).

  4. Patient who presents - barring the study disease - any previous or concurrent medical condition or any laboratory or clinical findings or any other condition that in the opinion of the investigator would be negatively affected by the study product or that would affect the study product or that precludes his participation, e.g. uncontrolled diabetes mellitus, adrenal insufficiency, cardiac impairment, repeated infections, metabolic alkalosis, chronic diarrhoea.

  5. Female patient who is pregnant or breast-feeding. 6. Patient who cannot stop potassium sparing diuretics (e.g. antagonists of aldosterone as such spironolactone, canrenoate and eplerenone, amiloride, triamterene), angiotensin converting enzyme inhibitors, angiotensin II receptor antagonists, tacrolimus, potassium desodic salts.

  7. Patient who received any medication that could interfere with the study treatment within 4 weeks before the inclusion in the study, including angiotensin converting enzyme inhibitors, angiotensin II receptor antagonists, tacrolimus, ciclosporine, potassium desodic salts,antibiotics.

  8. Patient who received potassium sparing diuretics 6 weeks before the inclusion in the study.

  9. Patient who presents contra indications to the administration of the study treatment such like known allergic reactions or hypersensitivity to the active pharmaceutical ingredients or other excipients of the formulations of the study treatment (such as lactose), history of difficult access to the oral administration route and/or conditions that may hamper compliance and/or absorption of the study treatment (e.g. any difficulty of swallowing, mal-absorption, delayed gastric emptying, oesophageal compression, intestinal obstruction or other chronic gastrointestinal disease).

  10. Patient who is admitted to hospital in emergency settings. 11. Patient who participated in a clinical trial within the last 3 months before enrolment.

  12. Patient who is at risk of non-compliance in the judgment of the investigator.

  13. Patient who could present any other condition, which in the opinion of the investigator, would preclude participation in the study.

  14. Patient who cannot be contacted in case of emergency. 15. Patient under any administrative or legal supervision.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of urinary pH values ≥ 7.0 during 24h on Day 7 (after ADV7103 treatment period) | 24 hours
  The primary endpoint is the comparison between the probability of having an urinary PH ≥ 7.0 based on all urinations during Day 7 in an ADV7103 dose versus the probability in the placebo group. All urinations on Day 7 with an evaluable pH measure will be included in the analysis. The study will be declared positive if the chance of having pH value ≥ 7.0 at each urination on D7 is superior with at least one ADV7103 treatment group than with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Luc-André Granier, Study Chair — Advicenne Pharma
Locations (12):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - UZ Leuven, Gasthuisberg Hospital, Leuven, Leuven
- France (10):
  - CHU Grenoble, Grenoble, Grenoble Cedex
  - CHRU Lille, Lille, Lille
  - CHU Pitié-Salpétrière, Paris, Paris
  - Hôpital Necker AP-HP, Paris, Paris
  - Hôpital Necker Enfants Malades, Paris, Paris
  - Hôpital Ténon - Explorations fonctionnelles Mutlidisciplinaires et INSERM UMR S 1155, Paris, Paris
  - Hôpital Américain CHU de Reims, Reims, Reims
  - CHU Reims, Reims, Reims
  - CHU Purpan, Toulouse, Toulouse Cedex 9
  - Centre Hospitalier Universitaire de Lyon - Hôpital Femme Mère Enfant, Bron

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website — http://advicenne.com/